CLINICAL TRIAL: NCT03908554
Title: The Effects of "Workplace Health Promotion Program" on Pain, Fatigue, Stress in Nurses: A Randomize Controlled Trail and One-Year Follow-up
Brief Title: The Effects of "Workplace Health Promotion Program" on Pain, Fatigue, Stress in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gokcen Akyurek, PhD PT, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 431-1271
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Nurses; Work-Related Stress Disorder; Pain; Fatigue
Keywords: coping skill; quality of life; pain; fatigue; Workplace Health Promotion Program
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: The WHPP was applied to the intervention group in the workplace for two times a week for five weeks. During the first 5 minutes of the session, breathing exercises, 20 minutes, PMR and 10 minutes, posture exercises were performed. PMR has progressed gradually to every session. The program is under control with a follow-up chart of what the participants do every day, and the participants were supported with various reminders (i.e., graphical leaflets on PMR techniques which also can be used as a guide while practicing at home). Participants of the control group rested in a room for 40 minutes and were told that they could read every session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The WHPP was applied to the intervention group in the workplace for two times a week for five weeks. During the first 5 minutes of the session, breathing exercises, 20 minutes, PMR and 10 minutes, posture exercises were performed. PMR has progressed gradually to every session. The program is under control with a follow-up chart of what the participants do every day, and the participants were supported with various reminders (i.e., graphical leaflets on PMR techniques which also can be used as a guide while practicing at home).
  Interventions: Other: WORKPLACE HEALTH PROMOTION PROGRAM
- Control (No Intervention): Participants of the control group rested in a room for 40 minutes and were told that they could read every session.

INTERVENTIONS:
Other: WORKPLACE HEALTH PROMOTION PROGRAM — WHPP was PMR training, posture and breath exercises, and ergonomic suggestions.
  Arms: intervention

SUMMARY:
Pain, fatigue, and stress lead to decrease on their work performance with biopsychosocial functioning disorders on nurses. This study was conducted to examine the effects of the "Workplace Health Promotion Program" (WHPP) on pain, fatigue, stress, professional quality of life (Pro-QoL) and coping skills for nurses.

DETAILED DESCRIPTION:
The investigators conducted a randomized control trail in 30 nurses admitted to their Hospital. Progressive relaxation training, posture and breath exercises and ergonomic suggestion as a WHPP was applied to the intervention group (n=15) during the five weeks. Visual Analogue Scale (VAS) was used to determine the pain, fatigue and stress levels of the nurses. Brief COPE and the Professional Quality of Life Scale, Version 4 (Pro-QoL) were used to evaluate the coping skills and quality of life. The evaluations were performed three times on all the participants as; before and after training and the one-year follow-up.

Inclusion criteria of this study were working actively and at least 40 hours working in a week. Participants who have psychiatric illnesses with or without medication, prior training or current use of relaxation therapy and participants without consent were excluded.

Eighty nurses aged between 18 and 65, working in a hospital have been informed about the study. Forty-three nurses who met the criteria and signed consent forms were included in this study. WHPP was PMR training, posture and breath exercises, and ergonomic suggestions.

ELIGIBILITY:
Inclusion Criteria:

* Working actively and at least 40 hours working in a week,
* Working as a nurse.

Exclusion Criteria:

* Have psychiatric illnesses with or without medication,
* Have prior training or current use of relaxation therapy and participants without consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Nurses
Enrollment: 30 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
The Professional Quality of Life Scale, Version 4 (ProQoL): | Change from Baseline to after 5 weeks and at a year
  ProQoL (has 30 items) measures the positive and negative effects experienced by those who choose to help people with pain and trauma (Stamm, 2009). It is made up of three subscales: Compassion Satisfaction (CS), Burnout, Secondary Traumatic Stress (STS). The ProQOL prompts participants to rate the frequency of the experience of certain feelings in their workplace with the clients in the last 30 days. Items are rated on a 6-point scale (from 0: never to 5:very often).
Coping Orientation to Problems Experienced (Brief COPE): | Change from Baseline to after 5 weeks and at a year
  Brief COPE (has 28 items) measures 14 different coping strategies and they targets three categories: problem-focused (active coping, planning, use of instrumental support), emotion-focused (use of emotional support, positive reframing, acceptance, religion, humor), and dysfunctional coping (venting, denial, substance use, behavioral disengagement, self-distraction, self-blame. Each statement is graded on a four-point Likert scale: 1 = very seldom, 2 = fairly seldom, 3
  = fairly often, 4 = very often.
Visual Analog Scale (VAS) | Change from Baseline to after 5 weeks and at a year
  VAS is a tool developed by Price et al., aims to measure subjective experience such as pain (Hasson & Arnetz, 2005). Also, in the literature, VAS was reported to have a better response(i.e., ability to detect clinically significant change) compared to the Likert scale and might also be more reliable and valid (Vickers, 1999). The scale was applied by marking a point on the vertical or horizontal line that corresponds to the severity of the pain/fatigue/stress felt by the person, with a length of 10 cm and two different names (0 = no pain, 10 = most severe pain). The distance between the marking point and the lowest tip of the line was measured in centimeters, and the numerical value found was indicative of the pain/fatigue/stress intensity of the person

IPD SHARING:
Plan to Share IPD: Undecided